CLINICAL TRIAL: NCT03791619
Title: Post-Approval Study of the TECNIS SYMFONY® Toric Lenses
Acronym: ANCORA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TIOL-205-STPA
Record Dates: First submitted 2018-12-11; First posted 2019-01-02 (Actual); Results first posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Cataract; Corneal Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Higher Cylinder Toric IOL (Active Comparator): Consented subjects that are eligible will have both eyes implanted with a TECNIS Symfony IOL. Each eye may have a different TECNIS Symfony IOL implanted, as determined by the surgeon and the TECNIS Symfony Toric IOL calculator; however, at least one eye must be implanted with either a Symfony Toric IOL Model ZXT150 (lower-cylinder group) or a Model ZXT300 or ZXT375 (higher-cylinder group) and the fellow eye must have the same or a lower toric power. The eye with the highest toric power IOL will determine the model group.
  Interventions: Device: Higher Cylinder Toric IOL
- Lower Cylinder Toric IOL (Active Comparator): Consented subjects that are eligible will have both eyes implanted with a TECNIS Symfony IOL. Each eye may have a different TECNIS Symfony IOL implanted, as determined by the surgeon and the TECNIS Symfony Toric IOL calculator; however, at least one eye must be implanted with either a Symfony Toric IOL Model ZXT150 (lower-cylinder group) or a Model ZXT300 or ZXT375 (higher-cylinder group) and the fellow eye must have the same or a lower toric power. The eye with the highest toric power IOL will determine the model group.
  Interventions: Device: Lower Cylinder Toric IOL

INTERVENTIONS:
Device: Higher Cylinder Toric IOL — Symfony Toric models ZXT300 and ZXT375 IOL
  Arms: Higher Cylinder Toric IOL
Device: Lower Cylinder Toric IOL — Symfony Toric model ZXT150 IOL
  Arms: Lower Cylinder Toric IOL

SUMMARY:
This study is a prospective, multicenter, bilateral, non-randomized, open-label, comparative, 6-month clinical study conducted at up to 50 sites in the USA.

ELIGIBILITY:
Inclusion Criteria:

* be at least 22 years old
* have cataracts in both eyes
* have a certain degree of astigmatism in at least one eye
* sign the written informed consent
* be willing and able to comply with examination procedures
* understand, read and write English to complete informed consent and questionnaires
* be available for study follow-up visits

Both eyes must qualify to be eligible to participate in the study

Exclusion Criteria:

* Currently participating in any other clinical study or have participated in a clinical study during the last 30 days
* Have a certain disease/illness such as poorly-controlled diabetes
* Have certain ocular conditions such as uncontrolled glaucoma
* Taking medication that may affect subject vision
* Have irregular corneal astigmatism
* Pregnant, plan to become pregnant during the study, or is breastfeeding

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision
Locations (23):
- United States (23):
  - Empire Eye & Laser Center, Bakersfield, California
  - Southern California Eye Physicians & Associates, Long Beach, California
  - Santa Monica Eye Medical Group, Santa Monica, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Florida Eye Microsurgical Institute, Inc., Boynton Beach, Florida
  - The Eye Associates of Manatee, Bradenton, Florida
  - Levenson Eye Associates, Jacksonville, Florida
  - North Florida Eye Surgeons, LLC dba Florida Eye Specialist, Jacksonville, Florida
  - Center For Sight, Sarasota, Florida
  - Virdi Eye Clinic & Laser Vision Care, Rock Island, Illinois
  - Chesapeake Eye Care & Laser, Annapolis, Maryland
  - Oakland Ophthalmic Surgery, Birmingham, Michigan
  - Tekwani Vision Center, St Louis, Missouri
  - Northern New Jersey Eye Institute PA, South Orange, New Jersey
  - Ludwick Eye Center, Chambersburg, Pennsylvania
  - Carolina Cataract & Laser Center, Ladson, South Carolina
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Memphis Eye & Cataract Associates, PLLC, Memphis, Tennessee
  - Cornea Associates of Texas, Dallas, Texas
  - Texas Eye & Laser Center, Hurst, Texas
  - Focal Point Vision, San Antonio, Texas
  - Parkhurst NuVision, San Antonio, Texas
  - Clarus Eye Centre, Lacey, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: It includes all subjects with ZXT300/375/150 toric IOL in the primary eye.
Groups:
- Higher Cylinder Group: All subjects implanted with a higher cylinder IOL (ZXT300 or ZXT375) in the primary eye.
- Lower Cylinder Group: All subjects implanted with a lower cylinder IOL (ZXT150) in the primary eye.
Period: Overall Study
Arm/Group | Higher Cylinder Group | Lower Cylinder Group
Started | 260 | 215
Completed | 256 | 209
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Population: Higher cylinder group consists of all subjects implanted with a higher cylinder IOL (ZXT300 or ZXT375) in the primary eye. Lower cylinder group consists of all subjects implanted with a lower cylinder IOL (ZXT150) in the primary eye.
Groups:
- Total: Total of all reporting groups
Arm/Group | Higher Cylinder Group | Lower Cylinder Group | Total
Number analyzed (Participants) | 260 | 215 | 475
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.2 (9.8) | 68.2 (7.9) | 68.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 134 | 285
  Male | 109 | 81 | 190
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 12 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 8 | 20
  White | 237 | 194 | 431
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Bothersome Visual Symptoms
Description: The rate of subjects reporting one or more of these items as very or extremely bothersome and impacting daily life via questionnaire.
Time Frame: 6-month
Population: Higher cylinder includes all bilaterally implanted subjects with at least a ZXT300 or ZXT375 in the primary eye; lower cylinder group includes all bilaterally implanted subjects with ZXT150 in the primary eye.
Measure: Count of Participants; unit: Participants
Arm/Group | Higher Cylinder Group | Lower Cylinder Group
Number analyzed (Participants) | 256 | 209
Participants | 19 | 19

2. Primary Outcome: Rate of Difficulty With an Activity Due to the Visual Symptoms
Description: The rate of reported difficulty with an activity due to one or more of visual symptoms impacting daily life via questionnaire.
Time Frame: 6-month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Higher Cylinder Group | Lower Cylinder Group
Number analyzed (Participants) | 256 | 209
Participants | 28 | 26

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Higher Cylinder Group | Lower Cylinder Group
All-Cause Mortality (participants affected / at risk) | 0/260 | 2/215
Serious Adverse Events (participants affected / at risk) | 34/260 | 33/215
Other Adverse Events (participants affected / at risk) | 12/260 | 2/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Higher Cylinder Group (N=260) | Lower Cylinder Group (N=215)
Cystoid Macular Edema (Eye disorders) | 7 (7) | 8 (10)
Vitreous Hemorrhage (Eye disorders) | 0 (0) | 1 (1)
Undesirable Optical Phenomena (Eye disorders) | 1 (1) | 2 (2)
Elevated IOP requiring treatment (Eye disorders) | 7 (8) | 7 (7)
Non-Ischemic Optic Neuropathy (Eye disorders) | 0 (0) | 1 (1)
Lens Axis Misalignment requiring SSI (Eye disorders) | 6 (6) | 0 (0)
Retinal Detachment/Tear (Eye disorders) | 1 (1) | 0 (0)
RETINAL VEIN OCCLUSION (Eye disorders) | 0 (0) | 1 (1)
Visual Symptoms requiring SSI (Eye disorders) | 2 (3) | 0 (0)
Tilt & decentration requiring SSI (Eye disorders) | 0 (0) | 1 (1)
IOP Elevated Without Need for Treatment (Eye disorders) | 3 (3) | 2 (2)
Corneal Edema (Eye disorders) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0)
IOP Greater than 10mmHg from Screening and More than 25mmHg (Eye disorders) | 0 (0) | 2 (2)
Hospitalization (General disorders) | 6 (8) | 5 (6)
Difficulty Breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cancer (General disorders) | 1 (1) | 1 (1)
Wrist Fracture Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Pneumonia/COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Higher Cylinder Group (N=260) | Lower Cylinder Group (N=215)
Undesirable Optical Phenomena (Eye disorders) | 12 (12) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communication prior to public release and can embargo communications regarding trial results at any time.

DOCUMENTS (2):
  • Study Protocol (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT03791619/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT03791619/SAP_001.pdf